CLINICAL TRIAL: NCT04360135
Title: Preemptive Acetaminophen for Postoperative Pain Control Following Minimally Invasive Hysterectomy: a Randomized Control Trial
Brief Title: Preemptive Acetaminophen for Postoperative Pain Control Following Minimally Invasive Hysterectomy
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was closed on 3/8/2021 as per final progress report issued by the IRB on 3/12/2021. No subjects were enrolled in the study following approval. Status changed to "Withdrawn (No Participants Enrolled)" accordingly.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-10702
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Preemptive acetominophen (Experimental): Acetaminophen 975mg BID the day before surgery and again 30-60 minutes preoperatively
  Interventions: Drug: Acetaminophen
- Standard of care (Placebo Comparator): Placebo the day before surgery and acetaminophen 30-60 minutes preoperatively
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Preemptive acetaminophen the day before surgery
  Arms: Preemptive acetominophen
Drug: Placebo — Preemptive placebo the day before surgery
  Arms: Standard of care

SUMMARY:
This study is investigating whether administration of acetaminophen the day before surgery improves post operative pain following minimally invasive hysterectomy. Patients will receive either acetaminophen or placebo to take twice per day the day prior to their scheduled surgery. The morning of surgery all participants will receive oral acetaminophen at least 30 minutes prior to surgery. The investigators will examine whether there is a difference in post operative pain between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing minimally invasive hysterectomy for benign indications

Exclusion Criteria:

* acetaminophen allergy
* liver disease
* kidney disease
* consume >3 alcoholic beverages per day
* weigh <50 kilograms
* report daily opiate use
* contraindication to acetaminophen
* used acetaminophen within 24 hours of surgery
* undergoing a concomitant pelvic reconstructive procedure

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Post-operative opioid use | 4 hours
  The total amount of opiate consumption in the immediate postoperative period will be recorded. Per standard protocol, patient's will be ordered for pain medication to receive on an as needed basis. The amount of both oral and IV opioids consumed by the patient will be converted to total morphine equivalents. As such, post operative opioid use will be used as a proxy for degree of post operative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Yettaw, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No